CLINICAL TRIAL: NCT03535688
Title: D-cycloserine for the Treatment of Chronic, Refractory Low Back Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding to complete the study
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00205398; A-20364 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-04-03; First posted 2018-05-24 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Pain
Keywords: Chronic Pain; Low Back Pain; D-cycloserine
MeSH Terms: conditions — Low Back Pain; Pain; Chronic Pain | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D-cycloserine (Experimental): D-cycloserine 200 mg twice daily
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 200 mg twice daily
  Arms: D-cycloserine
Drug: Placebo — twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of D-cycloserine versus placebo in relieving the signs and symptoms of patients with chronic lower back pain.

DETAILED DESCRIPTION:
This is a 26-week, double-blind, randomized, placebo-controlled two-arm parallel-group trial of d-cycloserine, a pharmacological treatment selected based on positive results from previous preclinical and clinical studies, for the treatment of chronic, refractory low back pain (CBP). After a 2-week screening period, individuals will be randomized to receive either 12 weeks of d-cycloserine or placebo and then followed for an additional 12 weeks to evaluate persistence of benefit at study endpoint, 24 weeks after randomization. During the 12-week treatment period, participants will undergo evaluation at baseline and at clinic visits on weeks 2, 6 and 12 after randomization to assess pain, proper treatment use and side effects. During the subsequent 12-week follow-up period, pain and safety will continue to be assessed monthly by phone calls. All patients will also be assessed daily using an electronic diary (eDiary) to record pain and mood. Magnetic resonance imaging (MRI), anatomical MRI, resting state functional MRI (fMRI), diffusion-tensor imaging (DTI) MRI, and arterial spin labeling (ASL) will be performed at baseline and at the end of 12 weeks for individuals completing MRI.

ELIGIBILITY:
Inclusion Criteria:

* Must have a history of low back pain for a minimum of 6 months with or without signs and symptoms of radiculopathy
* Male or female, age 18 years or older, (no racial/ethnic restrictions)
* Must have an average pain score of ≥ 4 (on a 0-10 NRS) over a 5-7 day period (minimum of daily eDiary entries for at least 5 of 7 days) immediately preceding the baseline visit (visit 2)
* Must be willing to read and able to understand instructions as well as patient reported outcomes (PROs)
* Must be in generally stable health
* Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate
* Must be willing to discontinue all pain medications for chronic back pain (listed below) except the study medication and rescue medication provided and not use the following prohibited pain medications throughout the duration of the treatment period

  * analgesics including over the counter (OTC) medications
  * NSAIDS including OTC medications
  * Coxibs
  * Opioids
  * Muscle relaxants
  * Gabapentins including pregabalin and gabapentin
* Must be willing to comply with recording pain, mood, and study treatment adherence twice daily using study eDiary
* Must be willing to abstain from drinking alcohol during the course of the study.
* If female, must be post-menopausal for at least one year or practicing an accepted, highly effective method of contraception or abstinence and plan to continue during the course of the study.

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, or history of surgery or tumor in the back within the past 6 months
* Involvement in litigation regarding their back pain or has a disability claim or is receiving workman's compensation or is seeking either as a result of their low back pain
* Epidural steroid injection within the past 3 months
* History of seizures
* Major new or untreated psychiatric disorder during the past 6 months and/or ongoing treatment with buproprion or fluphenazine
* Beck Depression Inventory II score of >28
* Significant renal disease or severe renal insufficiency
* Substance abuse/dependence including alcohol within the past 6 months
* Significantly abnormal laboratory values
* Pregnant or lactating at the time of randomization
* Known sensitivity to D-cycloserine
* Currently taking any of the following medications: ethionamide, dilantin, isoniazid (INH)
* In the judgment of the investigator, unable or unwilling to follow the protocol and instructions
* Any change in medication or physical therapy regime for back pain in the last 30 days.
* Chronic progressive neurologic conditions, including Parkinson's disease, Alzheimer's disease, and other conditions associated with dementia
* Other medical disease such as clinically significant congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy
* Presence of undiagnosed skin lesions or history of melanoma
* Current use of recreational drugs
* Current use of medical marijuana
* High dose opioid prophylaxis, defined as > 50mg morphine equivalent/day
* Intra-axial implants (e.g. spinal cord stimulators or pumps)
* Pregnancy or inability to use an effective method of birth control in sexually active men and women while taking the study drug and for one week thereafter. Barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUD's), hormonal contraceptives, oral contraceptive pills, surgical sterilization, and complete abstinence are examples of effective methods of contraception.
* Following laboratory abnormalities: liver function tests (SGOT/SGPT) greater than 2.5 times the upper limit of normal; unexplained anemia; evidence of renal insufficiency (creatinine > upper limit of normal) or any other abnormality that the principal investigator feels puts the participant at risk during the study.
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk
* Lactose allergy
* Ongoing participation in another clinical research study involving an investigational product or having received another investigational product within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) pain score 0-10; higher worse | 12 weeks
  Mean pain levels will be assessed at study baseline and compared to mean pain levels at Week 12 (study efficacy endpoint). Pain will be assessed using an 11-point NRS scale.

SECONDARY OUTCOMES:
Gender (male/female) | 12 weeks
  Assess the effect of gender on magnitude of pain response
Brain biomarkers (MRI) | 12 weeks
  Evaluate interaction between the primary endpoint and specified brain biomarkers, with particular attention to corticostriatal connectivity. Whole-brain exploratory analyses will also be used to identify both brain predictors or treatment response and brain reorganization in response to treatment.
Patient Global Assessment | 12 weeks
  A 5-point scale used to reflect the global impact of pain from the patient's perspective. Score 0-10; higher worse
Patient Global Impression of Change | 12 weeks
  A 7-point self-report measure that reflects a patient's belief about the efficacy of treatment; by depicting a patient's rating of overall improvement. Score 1-7, higher worse
McGill Pain Questionnaire (MPQ) | 12 weeks
  A 17-item self-reported measure assessing both the quality and intensity of subjective pain. Score 0-45, higher worse
PainDETECT Questionnaire (PDQ) | 12 weeks
  A 14-item self-reported measure assessing qualities for pain of neuropathic origin to distinguish pain severity. Score 0-38; higher more neuropathic
Beck Depression Inventory (BDI) | 12 week
  A 21-item self-report rating inventory that measures characteristic attitudes and symptoms of depression. Score 0-63, higher worse
Positive and Negative Affect Schedule (PANAS) | 12 weeks
  A self-report questionnaire consisting of two 10-item (5-point) scales to measure both positive and negative affects of pain. Score 10-50; higher more positive
Pain Catastrophizing Scale (PCS) | 12 weeks
  A 13-item scale assessing the degree of catastrophic cognitions in the sensation of pain.
  The scale ranges from 1 (not at all) to 4 (always). Score 0-52, higher worse
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 12 weeks
  A 32-item self-reported measure delineating between beneficial versus maladaptive interoceptive attention. Score 0-160, higher more awareness.
Oswestry Disability Index (ODI) | 12 weeks
  A 10-item self-reported measure quantifying a subjective percentage score of level of function (disability) in activities of daily living in those with chronic low back pain. Score 0-50; higher is greater disability
12-Item Short Form Survey (SF-12) | 12 weeks
  A 12-item self-report questionnaire measuring functional health and well-being from the patient's point of view. The SF-12 measures patient reported, health related quality of life from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Pinto CB, Bielefeld J, Barroso J, Yip B, Huang L, Schnitzer T, Apkarian AV. Chronic pain domains and their relationship to personality, abilities, and brain networks. Pain. 2023 Jan 1;164(1):59-71. doi: 10.1097/j.pain.0000000000002657. Epub 2022 Apr 20. No abstract available. PMID 35612403